CLINICAL TRIAL: NCT06813001
Title: Development of ACT (Acceptance and Commitment Therapy)-Based Nurse-led Intervention for Ovarian Cancer Patients
Brief Title: ACT-Based Nursing Intervention for Ovarian Cancer Patients: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2024-1286
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Neoplasm ; Psychological Distress
Keywords: Ovarian Neoplasms; Psychological Distress; Acceptand and Commitment Therapy (ACT); Nursing intervention
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental): Experimental group with application of ACT-based nursing intervention
  Interventions: Other: ACT-based nursing intervention

INTERVENTIONS:
Other: ACT-based nursing intervention — ACT-based nursing intervention is a 1:1 single online session with a nurse, which takes about 60 minutes followed by a daily self-monitoring survey for one week, which encourages patients to practice ACT.

SUMMARY:
The purpose of this study is to evaluate the feasiblity and effectiveness of an Acceptance and Commitment Therapy (ACT)-based nursing intervention aimed at managing psychological flexibility, distress, anxiety, depression, fear of cancer recurrence/progression, quality of life, and symptoms. Patients will participate in a single online session with a nurse, followed by a daily self-monitoring survey online for one week. Data will be collected at baseline (prior to the ACT session), on day 8 (after one week of self-monitoring), and at 5 weeks. Primary outcome is psychological flexibility.

DETAILED DESCRIPTION:
This study is a preliminary single-group pre-post design aimed at developing and evaluating the feasibility of an ACT-based nursing intervention for distress management in patients with ovarian cancer. A total of 25 ovarian cancer patients who consent to participate will be enrolled in the study. Paticipants will receive a one-time ACT-based nursing intervention lasting approximately 60 minutes.

The researcher will coordinate schedules with participants to deliver the ACT-based nursing intervention using Zoom, a video conferencing platform which minimizes time and location constraints. Before the intervention, the research will ensure that the participants' video conferencing is working properly to minimize potential difficulties during the session.

Following the single-session intervention, the researcher will send a daily Google Form link to participants for seven consecutive days. Participants will be encouraged to access the link and complete self-monitoring surveys to reinforce the key components addressed in the program.

ELIGIBILITY:
Inclusion Criteria:

* adult (19 ≤ age ≤ 75).
* ovarian cancer patients with FIGO stage 2-3.
* Those who have completed first-line chemotherapy for ovarian cancer (excluding maintenance therapy) within the past 2 years.

Exclusion Criteria:

* Patients with cognitive problems such as dementia or psychiatric problems such as major depression or generalized anxiety, or who are actively receiving treatment for any of these conditions.
* Patients with history of cancer recurrence.

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline psychological distress on the last day of self-monitoring (Day 8) | Psychological distress will be assessed at baseline and on the last day of self-monitoring (Day 8).
  Psychological distress measured by Distress Thermometer.

SECONDARY OUTCOMES:
Change from baseline depression | within 3 weeks after the last day of self-monitoring (window: 7 days)
  depression measured by the Hospital Anxiety and Depression Scale (HADS).
Change from anxiety | within 3 weeks after the last day of self-monitoring (window: 7 days)
  Anxiety by the Hospital Anxiety and Depression Scale (HADS).
Change from fear of cancer recurrence | within 3 weeks after the last day of self-monitoring (window: 7 days)
  Fear of cancer recurrence measured by the Fear of Cancer Recurrence Index (FCRI).
Change from psychological flexibility | within 3 weeks after the last day of self-monitoring (window: 7 days)
  Psychological flexibility measured by the Acceptance and Action Questionnaire-II (AAQ-II).
Change from quality of life | within 3 weeks after the last day of self-monitoring (window: 7 days)
  Quality of life measured by the ECORTC QLQ C-30.
Change from symptoms | within 3 weeks after the last day of self-monitoring (window: 7 days)
  Symptoms measured by the EORTC QLQ-OV28.

IPD SHARING:
Plan to Share IPD: No